CLINICAL TRIAL: NCT03136406
Title: NANT Pancreatic Cancer Vaccine: Combination Immunotherapy in Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-of-care Therapy
Brief Title: QUILT-3.039: NANT Pancreatic Cancer Vaccine: Combination Immunotherapy in Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-of-care Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.039
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide; Oxaliplatin; Capecitabine; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Bevacizumab; avelumab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT Pancreatic Cancer Vaccine (Experimental): A combination of agents will be administered to subjects in this study:
  cyclophosphamide, oxaliplatin, capecitabine, fluorouracil, leucovorin, nab-paclitaxel, bevacizumab, avelumab, ALT-803, aNK, GI-4000, and ETBX-011.
  Interventions: Drug: Cyclophosphamide; Drug: Oxaliplatin; Drug: Capecitabine; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: nab-paclitaxel; Biological: bevacizumab; Biological: avelumab; Biological: ALT-803; Biological: aNK for Infusion; Biological: ETBX-011; Biological: GI-4000

INTERVENTIONS:
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Oxaliplatin — cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: 5-Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
Drug: nab-paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
Biological: bevacizumab — Recombinant human anti-VEGF IgG1 monoclonal
Biological: avelumab — Recombinant human anti-PD-L1 IgG1 monoclonal antibody
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
Biological: aNK for Infusion — NK-92 cells
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with pancreatic cancer who have progressed on or after previous Standard of Care first line therapy and chemotherapy.

DETAILED DESCRIPTION:
Treatment will be administered in two phases. Subjects will continue treatment until they experience progressive disease (PD) or experience unacceptable toxicity (not correctable with dose reduction), withdraw consent, or the investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) will enter phase 2 of the study. Subjects may remain on phase 2 of the study for up to 1 year. Treatment will continue throughout phase 2 until the subject experiences PD or unacceptable toxicity, withdraws consent, or the investigator feels it is no longer in the subject's best interest to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
* Histologically-confirmed pancreatic cancer with progression on or after SoC therapy.
* ECOG performance status of 0 to 2.
* Have at least 1 measurable lesion and/or non-measurable disease evaluable according to RECIST Version 1.1.
* Must have a recent tumor biopsy specimen following the conclusion of the most recent anti-cancer treatment. If a historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period.
* Must be willing to provide blood samples for exploratory analyses.
* Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
* Agreement to practice effective contraception for female subjects with child-bearing potential and non-sterile males.

Exclusion Criteria:

* History of persistent grade 2 or higher (CTCAE Version 4.03) hematological toxicity resulting from previous therapy.
* History of other active malignancies or brain metastasis except: controlled basal cell carcinoma; prior history of in situ cancer (eg, breast, melanoma, cervical); prior history of prostate cancer that is not under active systemic treatment (except hormonal therapy) and with undetectable prostate-specific antigen (PSA) (< 0.2 ng/mL); bulky (≥ 1.5 cm) disease with metastasis in the central hilar area of the chest and involving the pulmonary vasculature. Subjects with a history of another malignancy must have > 5 years without evidence of disease.
* Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
* Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
* History of organ transplant requiring immunosuppression.
* History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
* Requires whole blood transfusion to meet eligibility criteria.
* Inadequate organ function, evidenced by the following laboratory results:

  * White blood cell (WBC) count < 3,500 cells/mm3
  * Absolute neutrophil count < 1,500 cells/mm3.
  * Platelet count < 100,000 cells/mm3.
  * Hemoglobin < 9 g/dL.
  * Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
  * Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
  * Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
  * Serum creatinine > 2.0 mg/dL or 177 μmol/L.
  * International normalized ratio (INR) or activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) >1.5 × ULN (unless on therapeutic anti-coagulation).
* Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
* Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
* Positive results of screening test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
* Known hypersensitivity to any component of the study medication(s).
* Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications. See Excluded Medications list.
* Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
* Concurrent participation in any interventional clinical trial.
* Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NANT Pancreatic Cancer Vaccine: A combination of agents will be administered to subjects in this study:
  cyclophosphamide, oxaliplatin, capecitabine, fluorouracil, leucovorin, nab-paclitaxel, bevacizumab, avelumab, ALT-803, aNK, GI-4000, and ETBX-011.
  Cyclophosphamide: 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Oxaliplatin: cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
  Capecitabine: 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
  5-Fluorouracil: 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Leucovorin: L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
  nab-paclitaxel: Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
  bevacizumab: Recombinant human anti-VEGF IgG1 monoclonal
  avelumab: Recombinant human anti-PD-L1 IgG1 monoclonal antibody
  ALT-803: Recombinant human super agonist interleukin-15 (IL-15) complex
  aNK for Infusion: NK-92 cells
  ETBX-011: Ad5 [E1-, E2b-]-CEA
  GI-4000: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
Period: Overall Study
Arm/Group | NANT Pancreatic Cancer Vaccine
Started | 3
Completed | 0
Not Completed | 3
Not completed — Treatment Discontinued-Investigator Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Histologically-confirmed pancreatic cancer with progression on or after SoC therapy. [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 30 days after last dose, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 30 days after last dose, up to 2 years or until resolution or stabilization for nonserious grade 3 or 4 AEs and SAEs, whichever is longer.
Arm/Group | NANT Pancreatic Cancer Vaccine
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=3)
Injection site erythema (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=3)
Neutropenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Injection site erythema (General disorders) | 3
Injection site reaction (General disorders) | 3
Pyrexia (General disorders) | 3
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Injection site pain (General disorders) | 1
Injection site swelling (General disorders) | 1
Pain (General disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Weight decreased (Injury, poisoning and procedural complications) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
INFUSION-RELATED REACTION - RIGORS (Investigations) | 1
Constipation (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Mucosal inflammation (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment. Only the safety data is provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT03136406/Prot_SAP_000.pdf